CLINICAL TRIAL: NCT06900348
Title: Prostate Specific Antigen Levels and Its Relationship With Some Characteristics in Individuals Living in Rural Areas: A Cross-Sectional Study
Brief Title: Prostate Specific Antigen Levels of Individuals Living in Rural Areas
Status: Not yet recruiting | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Feyza Bardak, Research Assistant, Suleyman Demirel University
Other Study IDs: TSTK-2024-9546; Suleyman Demirel Universty (Registry Identifier: TSTK-2024-9546)
Record Dates: First submitted 2025-03-22; First posted 2025-03-28 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Prostate Carcinoma
Keywords: Prostate Carcinoma, Screening
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: PSA-Activated PSA-PAH1 — Intravenous blood sample

SUMMARY:
It was planned in cross-sectional design in order to determine the specific prostate antigen level and some characteristics and the relationship evaluations and prostate specific antigen formation in individuals living in rural areas. It was planned to perform socio-demographic information formula, form including social information of health, prostate specific antigen test in the project data recording.

DETAILED DESCRIPTION:
It was planned in a cross-sectional design to evaluate the prostate specific antigen level and its relationship with some characteristics in elderly individuals living in rural areas and to determine the prostate specific antigen level. The research area of the project consists of 8 villages. In the collection of project data, it was planned to conduct a socio-demographic feature information form, a form including social determinants of health, and a prostate specific antigen test. This planned project is the first research to be conducted in our country in terms of determining risky groups, ensuring randomness in participants, and sampling method for universe representation. In addition, screening the rural area, which is disadvantaged in terms of socio-economic and demographic aspects, and preferring elderly individuals constitute the steps taken to ensure health equality of the disadvantaged group in terms of health service transportation opportunities.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 55 years or older

Exclusion Criteria:

-Prostate treatment

Min Age: 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male 55 years or older
Sampling Method: Probability Sample
Enrollment: 308 (Estimated)
Dates: Start 2025-03-25 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
PSA levels | 6 months
  For ages 60-69: 0 - 4.5 ng/ml, For ages 70 and above: 0 - 6.5 ng/ml

IPD SHARING:
Plan to Share IPD: No